CLINICAL TRIAL: NCT05734235
Title: Ultraviolet B Radiation-Induced Microvesicle Particle Release in Human Skin
Brief Title: UVB-Induced MVP Release in Human Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06201
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Ultraviolet B Radiation; Microvesicle Particles
MeSH Terms: interventions — Ascorbic Acid; Vitamin E

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin C & Vitamin E (Experimental): After subjects undergo UVB treatment then they will be instructed to take two Vitamin C and one Vitamin E tablets daily for 8 days.
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Vitamin C — Two Vitamin C tablets daily for 8 days.
Dietary Supplement: Vitamin E — One Vitamin E tablet daily for 8 days.

SUMMARY:
This study is designed to assess if ultraviolet B radiation (UVB) found in sunlight causes the release of microvesicle particles in human skin, and if antioxidant vitamins can block their production.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Ages 21 to 45
* Skin type: Fitzpatrick Type I or II

Exclusion Criteria:

* Have underlying diseases that could affect wound healing
* On medications that are known photosensitizers (e.g., doxycycline) or anti-inflammatories (e.g., NSAIDS [except for low-dose aspirin] or steroids)
* History of abnormal scarring (e.g., keloids)
* Should not be on Vitamin C or E supplements for past month
* Unable to understand/complete informed consent
* Large volar arm tattoos that would inhibit the ability to conduct/evaluate the skin testing
* Renal compromise/kidney stones or allergy to Vitamin C/Vitamin E or lidocaine anaesthetic
* Use of tanning bends or recent UVB exposure to the areas in the past 3 months
* Recent (within 1 week) use to sunscreen to volar forearms

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-03-05 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Change in microvesicle particles (MVP) levels from baseline | Day 8
  Levels of microvesicle particles will be determined from skin biopsies

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Wright State Physicians, Fairborn, Ohio, United States

DOCUMENTS (1):
  • Informed Consent Form (2021-12-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT05734235/ICF_000.pdf